CLINICAL TRIAL: NCT00114946
Title: A Randomized, Open-Label Trial Comparing Two Avastin (Bevacizumab)-Based Treatment Regimens for the First-Line Treatment of Metastatic Colorectal Cancer
Brief Title: A Study to Compare Two Avastin-Based Treatment Regimens for the Treatment of Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Purpose: Treatment
Other Study IDs: AVF3430n
Record Dates: First submitted 2005-06-20; First posted 2005-06-21 (Estimated); Last update posted 2006-05-29 (Estimated); Status verified 2006-05

CONDITIONS: Colorectal Cancer
Keywords: Metastatic Colorectal Cancer OASIS
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

INTERVENTIONS:
Drug: Avastin

SUMMARY:
This is a randomized, open-label, active-control, multicenter trial comparing two oxaliplatin/Avastin-based treatment sequences as first-line therapy for metastatic colorectal cancer. The study is designed to compare the efficacy of these two treatment sequences with respect to progression free survival (PFS) and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Metastatic or locally advanced and unresectable colorectal cancer
* Measurable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST)
* Age >= 18 years
* ECOG performance status of 0 or 1
* Adequate hematologic, hepatic, and renal function at the time of study entry to begin prescribed study therapy, according to institutional guidelines
* Use of an effective form of contraception during the study (for subjects of childbearing potential and their partners)

Exclusion Criteria:

* Prior treatment with Avastin
* Hypersensitivity to any of the study drugs or ingredients
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored Avastin cancer study
* History of any other malignancy (except squamous or basal cell carcinoma of the skin, carcinoma in situ of the cervix, or carcinoma in situ of the colon or rectum that has been effectively treated) unless in complete remission and off all therapy for that malignancy for at least 5 years
* Known brain or central nervous system metastases
* Prior treatment for advanced or metastatic colorectal cancer
* Prior treatment with an anti-angiogenesis agent, in either the adjuvant or metastatic setting
* Concurrent use of investigational anti-neoplastic agents (including up to 4 weeks prior to enrollment)
* Medical or psychiatric disorders that would interfere with informed consent or compliance, or would render the subject at high risk for participation in this study and its follow-up procedures
* Active infection requiring antibiotics on Day 1
* New York Heart Association (NYHA) Grade II or greater CHF
* Evidence of bleeding diathesis or coagulopathy
* Grade > 1 peripheral neuropathy (as defined by the NCI CTCAE, v3.0)
* Lack of physical integrity of the upper gastrointestinal tract or history of malabsorption syndrome
* Blood pressure > 150/100 mmHg
* Major surgical procedure, open biopsy, or significant traumatic injury within 30 days prior to Day 1; anticipation of need for a major surgical procedure during the course of the study
* Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to Day 1
* Urine protein:creatinine ratio >= 1.0 at screening
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 1
* Serious, non-healing wound, ulcer, or bone fracture
* History of myocardial infarction within 6 months prior to Day 1
* Unstable angina
* Clinically significant peripheral vascular disease
* History of stroke within 6 months prior to Day 1
* Pregnancy (positive pregnancy test) or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800
Dates: Start 2005-05; Study Completion 2007-12

PRIMARY OUTCOMES:
To compare the efficacy, as measured by progression-free survival (PFS), of FOLFOX/Avastin followed by FOLFIRI/Avastin versus FOLFOX/Avastin followed by 5-FU/LV/Avastin as first-line therapy for previously untreated metastatic colorectal cancer.

SECONDARY OUTCOMES:
To evaluate the tolerability of sequential treatment in subjects and to evaluate the safety of an irinotecan/Avastin-based regimen versus a 5-FU/Avastin regimen for previously untreated metastatic colorectal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Sugrue, M.D., Study Director — Genentech, Inc.